CLINICAL TRIAL: NCT00975104
Title: A Randomized, Double-blind, Placebo-controlled Dose Ranging Study to Evaluate the Safety and Efficacy of AMG 745 in Age-associated Muscle Loss
Brief Title: AMG 745 in Subjects With Age-associated Muscle Loss
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Amgen has chosen at this time not to continue with AMG 745 study 20080733
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080733
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Age-associated Muscle Loss
Keywords: Aging; Frailty; Sedentary; Immobilization; Atrophy; Muscle Wasting; Physical Activity
MeSH Terms: conditions — Frailty; Sedentary Behavior; Atrophy; Muscular Atrophy; Motor Activity | interventions — AMG 745

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- AMG 745 0.3 mg/kg (Experimental): 0.3 mg/kg AMG 745
  Interventions: Drug: AMG 745 0.3 mg/kg
- AMG 745 1.0 mg/kg (Experimental): 1.0 mg/kg, AMG 745
  Interventions: Drug: AMG 745 1.0 mg/kg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- AMG 745 3.0 mg/kg (Experimental): 3.0 mg/kg, AMG 745
  Interventions: Drug: AMG 745 3.0 mg/kg

INTERVENTIONS:
Drug: AMG 745 0.3 mg/kg — AMG 745 0.3 mg/kg IV QW
  Arms: AMG 745 0.3 mg/kg
Drug: AMG 745 1.0 mg/kg — AMG 745 1.0 mg/kg IV QW
  Arms: AMG 745 1.0 mg/kg
Drug: AMG 745 3.0 mg/kg — AMG 745 3.0 mg/kg IV QW
  Arms: AMG 745 3.0 mg/kg
Drug: Placebo — Placebo IV QW
  Arms: Placebo

SUMMARY:
Randomized, Double-blind, Placebo-controlled Dose Ranging Study to Evaluate the Safety and Efficacy of AMG 745 in Age-associated Muscle Loss

ELIGIBILITY:
Inclusion Criteria:

* Limited exercise tolerance and Rapid Assessment of Physical Activity (RAPA) score ≤ 3
* Hand grip (dominant hand): men ≤ 30.3 kg, women ≤ 19.3 kg
* Walk speed ≤ 0.8 m/s (based on a 4 meter walk)

Exclusion Criteria:

* Subject weight > 137 kg (300 lbs), or Body Mass Index (BMI) > 32 kg/m2
* Primary muscle disease or myopathy
* Recent immobilization, or major trauma to the legs within 6 months
* Knee or hip replacement within 12 months or lower extremity amputation
* Significant laboratory abnormalities
* Significant comorbidities or medical history
* Weight loss (intentional or unintentional) of > 5 kg in 12 weeks
* Unable to complete an MRI scan

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of AMG 745 weekly IV doses of 0.3 mg/kg, 1.0 mg/kg, or 3.0 mg/kg, compared with weekly IV placebo on thigh muscle CSA in subjects ≥ 65 yrs old with limited exercise tolerance and functional limitations | 12 Weeks

SECONDARY OUTCOMES:
To evaluate the effect of treatment with AMG 745 on muscle strength (hand grip strength) and function (gait speed, 10-step stair climb power, chair stand and 6 minute walk distance) and to evaluate the PK of AMG 745 following multiple IV administrations | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com